CLINICAL TRIAL: NCT04747444
Title: The Effects of Anti-Gravity Treadmill Walking In Individuals With Knee Osteoarthritis
Brief Title: Positive Pressure Treadmill Walking for Individuals With Knee Pathology
Acronym: LBPPKNEEOA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Prakash Jayabalan MD, PhD, Principle Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 00209531
Record Dates: First submitted 2020-12-11; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Individuals with knee osteoarthritis will walk 45 minutes on a treadmill at 100% full body weight loading
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100% body weight walking (Other): Individuals with knee osteoarthritis will walk 45 minutes on a treadmill at 100% full body weight loading
  Interventions: Other: Anti-Gravity Treadmill
- 50% body weight walking (Other): Individuals with knee osteoarthritis will walk 45 minutes on a treadmill at 50% full body weight loading
  Interventions: Other: Anti-Gravity Treadmill

INTERVENTIONS:
Other: Anti-Gravity Treadmill — Treadmill in which the body weight percent placed on the lower extremities can be controlled

SUMMARY:
Our goal is to compare the serum biomarker changes of joint disease that occur in response to partially off-loaded (50%) walking exercise to regular (100%) walking exercise while on a Lower Body Positive Pressure (LBPP) treadmill. Secondly we are determining the relationship between changes in the concentration of these serum biomarkers and participant reported knee pain while walking on a LBPP treadmill.

DETAILED DESCRIPTION:
The morphology and composition of healthy mature articular cartilage is optimized to its primary function of load transfer and distribution. In the osteoarthritic state however, homeostasis of the knee joint is significantly altered, such that as load is placed on the joint there is progressive worsening of cartilage damage over time. Altered joint mechanics and intra-articular biological processes are thought to play pivotal roles in the initial breakdown and potentiation of cartilage damage which is the hallmark finding in knee OA leading to knee pain. Walking or running with weight support on a lower-body positive-pressure (LBPP) treadmill is a novel training and rehabilitation modality for individuals with lower extremity pathologies due to its ability to limit pain. This treadmill provides a controlled off-loading of the lower extremities with significant benefit being shown after 12 weeks of training in overweight individuals with knee OA on knee pain, function and muscle strength. Although this methodology alters the joint mechanics, the intra-articular biological effect on joint disease remains unknown.

A recent study from our laboratory compared walking exercise on a regular treadmill at a defined speed with and without rest breaks in 27 participants with knee OA and demonstrated that one-hour rest breaks had significant benefits. This conclusion was based on reduction in knee joint contact force and decreased levels of a serum marker commonly associated with cartilage degradation (cartilage oligomeric matrix protein, COMP) at 45 minutes of walking. This investigation assessed patterns of walking, but the impact of varying knee joint contact force, such as by walking on a LBPP treadmill on the biological profiles of joint disease is not known. The present study will establish the conditions and parameters for a future longer-term clinical trial that aims to individualize the amount of joint loading during LBPP treadmill training in participants with knee OA based on their biomarker profile.

Objective 1: Compare the serum biomarker changes of joint disease that occur in response to partially off-loaded (50%) walking exercise to regular (100%) walking exercise while on a LBPP treadmill.

Objective 2: Determine the relationship between changes in the concentration of these serum biomarkers and participant reported knee pain while walking on a LBPP treadmill.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Diagnosis of unilateral or bilateral knee osteoarthritis
* Clinical AND/OR radiographic knee osteoarthritis.

Exclusion Criteria:

* Age < 50 years
* History of lower extremity total joint arthroplasty
* Current cardiovascular disease or hypertension that is uncontrolled
* History of neurological disorder that effects lower extremity function (i.e., stroke, peripheral neuropathy, multiple sclerosis, Parkinson's disease)
* Current ankle or hip pain
* Currently pregnant for female participants
* Weight over 400 lbs (181.4 kg), height less than 4'8" (142 cm) or over 6'4" (193 cm), 18.5" (47 cm) hip width, or 58" (147 cm) hip circumference

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in Cartilage oligomeric matrix protein serum concentration | baseline, and 45 minutes of walking
  Serum (blood) marker concentration
Change in Knee Joint Pain | baseline, and 45 minutes of walking
  Numeric pain rating scale (NPRS). Higher scores on this scale indicate higher pain

SECONDARY OUTCOMES:
Change in Inflammatory cytokine (IL-6, IL-1B and TNF-A) concentration | baseline, and 45 minutes of walking
  Serum (blood) marker concentration

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Jayabalan, MD, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No